CLINICAL TRIAL: NCT06084221
Title: Fatal Overdose Review Teams - Research to Enhance Surveillance Systems (FORTRESS)
Brief Title: Fatal Overdose Review Teams - Research to Enhance Surveillance Systems
Acronym: FORTRESS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Matthew Aalsma, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15922; 1R61DA057660-01 (NIH); 4R33DA057660-02 (NIH)
Record Dates: First submitted 2023-09-25; First posted 2023-10-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Substance-Related Disorders; Opioid-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFR Team Practice as Usual (No Intervention): Data are collected regarding standard OFR Team practice and outcomes before implementation of the FORTRESS Intervention
- FORTRESS (Experimental): Participating counties receive both training in data-driven decision making and inventory of overdose-prevention strategies
  Interventions: Behavioral: Data-Driven Decision Making (DDDM); Behavioral: Overdose-prevention strategies inventory

INTERVENTIONS:
Behavioral: Data-Driven Decision Making (DDDM) — The intervention consists of providing real-time data on overdose touchpoints to OFRs and training in DDDM for continuous quality improvement cycles, leading to improved OFR recommendations and implementation of overdose prevention strategies.
  Arms: FORTRESS
Behavioral: Overdose-prevention strategies inventory — A list of overdose prevention and harm reduction strategies will be provided to OFRs for possible implementation, depending on local needs and final dashboard development.
  Arms: FORTRESS

SUMMARY:
This project seeks to address the overdose epidemic by working with overdose fatality review (OFR) teams. Current OFR practices rely on a case review model where OFR teams assess one or two overdose cases to make policy and program recommendations. However, the continued rise in overdose rates and number of preventable overdose deaths suggest a need to shift OFR teams away from case review and toward using timely population-level data to better inform their recommendations and actions.

The goal of this project, Fatal Overdose Review Teams - Research to Enhance Surveillance Systems (FORTRESS), is to improve standard OFR practices by equipping OFRs with a data dashboard built on near real-time aggregate data, linked across multiple sources and presented in a way that helps identify common "overdose touchpoints," or opportunities to connect individuals at risk for overdose with evidence-based treatment.

During the first project phase, the FORTRESS team will design the "Overdose Touchpoints Dashboard'' (Aim 1). The FORTRESS team will also train OFR team members in "Data-Driven Decision Making" (DDDM) to effectively use the dashboard. The FORTRESS team also includes individuals involved in developing the CDC's OFR best practice guidelines and a pilot study of OFR adherence to these guidelines, which will inform the FORTRESS team's development of an "OFR Fidelity Tool'' (Aim 2). This tool will be the first of its kind.

For the second project phase, the FORTRESS team will conduct a cluster-randomized stepped-wedge trial comparing the impact of the intervention (dashboard + DDDM training) versus standard OFR practices on both implementation (Aim 3) and effectiveness outcomes (Aim 4). Implementation outcomes include implementation process fidelity (Stages of Implementation Completion), staff acceptance of harm reduction philosophies (qualitative interviews), OFR fidelity to CDC best practices (FORTRESS OFR Fidelity Tool), and usability of the Overdose Touchpoint Dashboard, (Systems Usability Scale). A statewide OFR data repository serves as a rich source of data on effectiveness outcomes, including OFR team recommendation quality and local actions to implement recommended overdose prevention strategies. The FORTRESS team will also survey OFR team members to assess changes in their attitudes toward evidence-based overdose prevention strategies. In sum, the FORTRESS team is uniquely qualified to help OFRs use more comprehensive available data to inform quality, action-oriented recommendations to reduce overdose. Funding for this project comes from the HEAL Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria for FORTRESS staff personnel recruited to complete surveys, focus groups and/or interviews:

* 1) member of local overdose fatality review (OFR) team; OR 2) local county leader of organizations represented by OFR (OFR facilitator, public jail administrators, chief of police, judge, addiction treatment CEO/CFO, public health director, etc.).

Inclusion criteria for FORTRESS administrative data:

* all residents of Indiana that have experienced fatal and/or non-fatal overdose as identified by administrative data sources.

Exclusion Criteria

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Organizational readiness to implement change | Months 18, 24, 30, 36, 42, 48, 54, & 60
  12-items that assess perceived readiness to implement new innovations that will be administered to 15 OFR team members and 5 system leaders per each of 18 counties.
Cultural Exchange Inventory (adapted to evaluate OFR team alliance) | Months 18, 24, 30, 36, 42, 48, 54, & 60
  15-items that measure knowledge and attitudes between organizations that will be administered to 15 OFR team members and 5 system leaders per each of 18 counties.
Harm reduction acceptability scale | Months 18, 24, 30, 36, 42, 48, 54, & 60
  25-items that measures the adoption of a harm reduction approach in responding to people who use substances that will be administered to 15 OFR team members and 5 system leaders per each of 18 counties.
Systems Usability Scale | Months 18, 24, 30, 36, 42, 48, 54, & 60
  10-items that assesses the usability of dashboard for OFRs that will be administered to 15 OFR team members and 5 system leaders per each of 18 counties.
Stages of Implementation Completion (SIC) | Baseline through study completion, an average of 5 years
  The SIC is a measure of implementation process fidelity and allows for continuous measurement of implementation success. The SIC is an observation-based assessment tool that qualitatively measures intervention implementation process and fidelity. Assessment of the SIC results will be ongoing across the intervention time period and into sustainment.
OFR Fidelity Tool | Months 18-54
  To be developed fidelity assessment tool that will be completed by each OFR facilitator after a monthly meeting.
Dashboard Aggregate Usage | Months 14-54
  Web Cookies and anonymized IDs for each unique user to track dashboard usage that will be tracked on an on-going basis. Dr. Reda will review results monthly.
Organization's implementation climate (adapted to evaluate overdose prevention strategies) | Months 18, 24, 30, 36, 42, 48, 54, & 60
  18-items that assesses the degree to which the climate is supportive of adopting new innovations that will be administered to 15 OFR team members and 5 system leaders per each of 18 counties.
Quality OFR Recommendations | Months 14-54
  OFR team recommendations will be gathered monthly. We will be coding the quality of OFR team recommendations using the coding system that we developed in phase 1 of our FORTRESS project. This measure involves qualitative assessments of whether a recommendation meets certain standards of quality. The qualitative coding will be conducted by research staff in a digital spreadsheet.
Uptake of OFR Interventions | Months 14-54
  OFR team recommendations will be gathered monthly. Uptake of an intervention will be defined as implementation of the recommendation. OFR team overdose prevention recommendations will be coded for uptake (whether or not they were implemented). This measure involves quantitative assessment of the incidence of uptake.
Overdose | Month 35-40 (interim) and month 53-57 (final)
  Mortality data is collected via death certificates that are submitted by county coroners to the IDOH Division of Vital Records, which include information on underlying cause of Death. Data will include all fatal accidental drug overdose deaths (X40-X44).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Aalsma, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States